CLINICAL TRIAL: NCT02593617
Title: The Effect of Energy Drink Consumption on Alcohol-Substance Use and It's Relationship With Impulsivity In University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafakemalpasa State Hospital (Other)
Responsible Party: Principal Investigator, Nil Banu Bahadırlı, Specialist, Mustafakemalpasa State Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: TUTF-GOKAEK 2012/196
Record Dates: First submitted 2015-10-29; First posted 2015-11-02 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Energy Drinks; Alcohol Drinking; Substance Use; University Students
Keywords: Energy Drinks; Alcohol Drinking; Substance Use
MeSH Terms: conditions — Alcohol Drinking; Substance-Related Disorders | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- University students who use alcohol (Other): In Addiction Profile Index, university students who use alcohol in last year.
  Interventions: Other: Addiction Profile Index; Other: Alcohol Use Disorders Identification Test; Other: Barratt Impulsiveness Scale; Other: Zuckerman Sensation Seeking Scale; Other: Energy Drink Consumption Questionnaire
- University students who don't use alcohol (Other): In Addiction Profile Index, university students who don't use alcohol in last year.
  Interventions: Other: Addiction Profile Index; Other: Alcohol Use Disorders Identification Test; Other: Barratt Impulsiveness Scale; Other: Zuckerman Sensation Seeking Scale; Other: Energy Drink Consumption Questionnaire
- University students who use energy drinks (Other): In energy drink consumption questionnaire, university students who use energy drinks in last year.
  Interventions: Other: Addiction Profile Index; Other: Alcohol Use Disorders Identification Test; Other: Barratt Impulsiveness Scale; Other: Zuckerman Sensation Seeking Scale; Other: Energy Drink Consumption Questionnaire
- University students who don't use energy drinks (Other): In energy drink consumption questionnaire, university students who don't use energy drinks in last year.
  Interventions: Other: Addiction Profile Index; Other: Alcohol Use Disorders Identification Test; Other: Barratt Impulsiveness Scale; Other: Zuckerman Sensation Seeking Scale; Other: Energy Drink Consumption Questionnaire
- University students who use substance (Other): In Addiction Profile Index, university students who use substance in last year.
  Interventions: Other: Addiction Profile Index; Other: Alcohol Use Disorders Identification Test; Other: Barratt Impulsiveness Scale; Other: Zuckerman Sensation Seeking Scale; Other: Energy Drink Consumption Questionnaire
- University students who don't use substance (Other): In Addiction Profile Index, university students who don't use substance in last year.
  Interventions: Other: Addiction Profile Index; Other: Alcohol Use Disorders Identification Test; Other: Barratt Impulsiveness Scale; Other: Zuckerman Sensation Seeking Scale; Other: Energy Drink Consumption Questionnaire

INTERVENTIONS:
Other: Addiction Profile Index
Other: Alcohol Use Disorders Identification Test
Other: Barratt Impulsiveness Scale
Other: Zuckerman Sensation Seeking Scale
Other: Energy Drink Consumption Questionnaire

SUMMARY:
The objective of this study is to investigate the prevalence of energy drink, alcohol and substance use among university students; to explore whether there is a relationship between energy drink consumption and alcohol-substance use in university students or not and to evaluate effect of impulsiveness and sensation seeking on this relationship.

ELIGIBILITY:
Inclusion Criteria:

* To be university student
* To be ≥ 18 years old

Exclusion Criteria:

* Not willing to participate the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2623 (Actual)
Dates: Start 2012-12; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Measurement of the prevalence of energy drink consumption among university students by using energy drink consumption questionnaire | One hour
Measurement of the prevalence of alcohol consumption among university students by using addiction profile index | One hour
Measurement of the prevalence of substance use among university students by using addiction profile index | One hour
Assessment of sensation seeking among university students by using Zuckerman Sensation Seeking Scale | One hour
Assessment of impulsivity among university students by using Barratt Impulsiveness Scale | One hour

CONTACTS AND LOCATIONS:
Locations (1):
- Mustafakemalpasa State Hospital, Bursa, Turkey (Türkiye)

REFERENCES:
- [Result] Arria AM, Caldeira KM, Kasperski SJ, Vincent KB, Griffiths RR, O'Grady KE. Energy drink consumption and increased risk for alcohol dependence. Alcohol Clin Exp Res. 2011 Feb;35(2):365-75. doi: 10.1111/j.1530-0277.2010.01352.x. Epub 2010 Nov 12. PMID 21073486
- [Result] Brache K, Stockwell T. Drinking patterns and risk behaviors associated with combined alcohol and energy drink consumption in college drinkers. Addict Behav. 2011 Dec;36(12):1133-40. doi: 10.1016/j.addbeh.2011.07.003. Epub 2011 Jul 23. PMID 21840130
- [Result] Marczinski CA. Alcohol mixed with energy drinks: consumption patterns and motivations for use in U.S. college students. Int J Environ Res Public Health. 2011 Aug;8(8):3232-45. doi: 10.3390/ijerph8083232. Epub 2011 Aug 5. PMID 21909303
- [Result] Velazquez CE, Poulos NS, Latimer LA, Pasch KE. Associations between energy drink consumption and alcohol use behaviors among college students. Drug Alcohol Depend. 2012 Jun 1;123(1-3):167-72. doi: 10.1016/j.drugalcdep.2011.11.006. Epub 2011 Dec 3. PMID 22138539